CLINICAL TRIAL: NCT02568475
Title: Involving Nursing Home Residents and Their Families in Acute Transfer Decisions: Pilot Test of a New Decision Aid
Brief Title: Involving Nursing Home Residents and Their Families in Acute Care Transfer Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Responsible Party: Principal Investigator, Ruth Tappen, Christine E. Lynn Eminent Scholar and Professor, Florida Atlantic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 343268; 1IP2PI000281-01 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Chronic Disease; Acute Disease
Keywords: nursing home residents, decision aid, acute care transfers
MeSH Terms: conditions — Chronic Disease; Acute Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision aid (Experimental): Provision of "Go to the Hospital or Stay Here?"
  Interventions: Behavioral: Provision of "Go to the Hospital or Stay Here?"
- No decision aid (No Intervention): Does not receive the decision aid.

INTERVENTIONS:
Behavioral: Provision of "Go to the Hospital or Stay Here?" — Residents and families randomly assigned to the intervention group (one half of the residents and one half of the families enrolled) are given the new Decision Aid to review with an RA trained for this purpose by the investigators. The Decision Aid provides information on risks and benefits of acute care transfer and information on advance care planning, resident and families' right to be involved in the decision. Resident or family member is also asked to re-read it and think about it over the subsequent 14 days.
  Other Names: Transfer Decision Guide
  Arms: Decision aid

SUMMARY:
This study addresses the Patient-Centered Outcomes Research Institute (PCORI) area of interest related to development of decision support tools that bring patients, families and clinicians together to decide, in this instance, whether or not transfer from the nursing home (NH) to acute care is necessary and appropriate. The purposes of this study were 1) to develop an evidence-based decision aid addressing potentially avoidable transfers of residents from nursing homes to hospitals (preceded this protocol), and 2) to evaluate this decision aid in terms of acceptability to residents and families and its effect on the quality of transfer decisions.

The primary hypotheses to be tested are:

Hypothesis 1: Resident and family members in the intervention group will report greater preparation for decision making and less decisional conflict than those in the no treatment control group.

Hypothesis 2: Residents and family members in the intervention group will demonstrate increased knowledge related to acute care transfer and less preference for acute care transfer than those in the no treatment control group.

DETAILED DESCRIPTION:
Project Summary: The goal of this project is to develop (Phase I) and test (Phase II) a new Transfer Decision aid that will better prepare nursing home (NH) residents and their families to participate in decisions to transfer the resident to an acute care facility or remain in the NH for treatment.

Objectives: The specific aim of this study is to evaluate the decision aid, "Go to the Hospital or Stay Here?" in terms of acceptability to residents and families and its effect on decision making and transfer decisions by residents and families.

Study Design: A mixed methods design was used to address the study aims. In Phase I (not submitted to ClinicalTrials.gov), interviews of a diverse sample of NH residents, their family members, primary care providers, nurses and social workers in the NH were conducted and the results were used to create a Transfer Decision aid to be pilot tested in Phase II for its effect on decision making and transfer decisions.

Phase II involves a pretest, intervention for the half randomly selected to receive it, 14 day posttest and 90 day follow-up.

Study Population: Staff of 15 participating South Florida nursing homes (NHs) were asked to recommend residents and family members of residents who could participate in the study. Residents were tested for ability to provide consent using the Mini-Cog prior to enrollment.

General Analytic Strategy: Multiple linear regression (MLR) will be used to analyze the variance when predicting the primary and secondary outcome variables, preparation for decision making, decisional conflict, knowledge and number of transfers (McNeil, Newman & Kellee, 1996; Pedhazur & Schmelking, 1991). For qualitative data, Phase II interviews are transcribed and the transcriptions reviewed for accuracy. Responses were de-identified (names, gender and ethnic identity information removed). A framework for descriptive (labeling and categorizing), interpretive (based on underlying meaning) and pattern (thematic) codes was developed. Intercoder reliability was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult nursing home resident and/or family member or identified significant other of a nursing home resident. Cognitively unimpaired individuals. Long or short term residents of nursing home or rehabilitation center.

Exclusion Criteria:

* Dementia as indicated by score on Mini-Cog. Inability to respond to questions due to physical disability or illness.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth M. Tappen, EdD, RN, FAAN, Principal Investigator — Christine E. Lynn College of Nursing, Florida Atlantic University
Locations (1):
- Florida Atlantic University, Christine E. Lynn College of Nursing, Boca Raton, Florida, United States

REFERENCES:
- [Result] Tappen RM, Worch SM, Elkins D, Hain DJ, Moffa CM, Sullivan G. Remaining in the nursing home versus transfer to acute care: resident, family, and staff preferences. J Gerontol Nurs. 2014 Oct;40(10):48-57. doi: 10.3928/00989134-20140807-01. PMID 25275783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decision Aid | No Decision Aid
Started | 97 | 95
Post-test | 85 | 82
Completed (3 month follow-up) | 46 | 52
Not Completed | 51 | 43
Not completed — Lost to Follow-up | 40 | 39
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Discharged home | 4 | 4
Not completed — Short-term: Discharge location unknown | 4 | 0
Not completed — Transferred to another facility | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid | No Decision Aid | Total
Number analyzed (Participants) | 97 | 95 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 12 | 31
  >=65 years | 78 | 83 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.69 (12.72) | 79.3 (13.94) | 78.05 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 63 | 129
  Male | 31 | 32 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 93 | 86 | 179
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 20 | 25
  White | 87 | 74 | 161
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Southeast Florida | 97 | 95 | 192
  United States: Elsewhere | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Preparation for Decision Making
Description: Range of possible raw scores: 10 - 50. Items can be summed and scored (sum the 10 items and divide by 10).
  There are no subscales. A higher score is positive indicating perception of being better prepared to make the decision identified when test is administered.
Time Frame: Decision Aid group only: Post test (2-3 weeks after pretest) and at 3 month follow-up (after post test)
Population: This analysis only included those that received the Decision Aid intervention and were collected at the end of the intervention (Time Point 2) and with a 3-month follow-up. Only 39 participants were still residents in the nursing homes during the 3-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Decision Aid: Received and Discussed the Decision Aid
  Provision of "Go to the Hospital or Stay Here?": Residents and families randomly assigned to the intervention group (one half of the residents and one half of the families enrolled) are given the new Decision Aid to review with an RA trained for this purpose by the investigators. The Decision Aid provides information on risks and benefits of acute care transfer and information on advance care planning, resident and families' right to be involved in the decision. Resident or family member is also asked to re-read it and think about it over the subsequent 14 days.
Arm/Group | Decision Aid | No Decision Aid
Number analyzed (Participants) | 39 | 0
score on a scale
  Post test | 39.59 (9.113) |
  3 month follow-up | 36.00 (10.084) |
Statistical Analysis 1: Comparison: Decision Aid; Test type: Equivalence — Continuous scale: score compares results before and after intervention without a cut parameter; p = 0.046, t-test, 2 sided; Mean Difference (Final Values) = 3.59, 95% CI 2-sided [0.059 to 7.12], Standard Error of Mean 1.74

2. Primary Outcome: Decisional Conflict Scale
Description: Scale Range of possible raw scores: 0 - 64.
  A lower score indicates less decisional conflict related to making the identified decision. Decisional conflict is a state of uncertainty about a course of action. Decision supporting interventions are thought to be effective in
Time Frame: Decision aid: Pretest (baseline) and Post test (2-3 weeks after pretest); No decision aid: Post test only
Population: Nursing Home Residents and Family Members. Only data for the Decision Aid group was collected for this outcome. The No Decision Aid Group, didn't receive the intervention and no data was analyzed before pre-test, therefore no data was collected. However, the score was analyzed in the No Decision Aid group (N=78) at the post-test time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Aid | No Decision Aid
Number analyzed (Participants) | 84 | 78
score on a scale
  Pretest | 13.11 (12.01) | NA (NA) — The No Decision Aid group did not do the Decision Aid during Pretest
  Post test | 9.39 (9.98) | 15.73 (14.68)
Statistical Analysis 1: Comparison: Decision Aid vs No Decision Aid; Test type: Other — This is a continuous scale with no clinical cut score/value. We tested mean differences between the two groups; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 6.78, 95% CI 2-sided [2.9 to 10.6]

3. Secondary Outcome: Knowledge Test
Description: Decision Aid Quiz Investigator Developed: True/False Test of Knowledge based upon information in the Decision Aid.
  Scale Range: 0 - 22. Total score is the number of questions answered correct.
  A higher score indicates greater number of responses are correct. Items are scored as 0 = incorrect; 1 = correct.
  Criteria used to assess this measure:
  Items based upon concept mapping of the Decision Aid Reviewed by a panel of experts prior to administration
Time Frame: Pretest (baseline) and Post test (2-3 weeks after pretest)
Population: Nursing Home Residents and Family Members
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Aid | No Decision Aid
Number analyzed (Participants) | 82 | 79
score on a scale
  Pretest | 15.63 (2.69) | 15.19 (2.64)
  Post test | 17.38 (2.86) | 15.80 (2.56)

4. Secondary Outcome: Treatment Preference/Decisional Conflict Scale
Description: Treatment Site Option Preference Administered prior to the Decisional Conflict Scale, this single item was used to ask participants if they preferred treatment in the hospital or nursing home or if the preference depended upon the seriousness of their condition (three choices). This is nominal level data. The administration of the item precedes administration of the Decisional Conflict Scale (DCS) described previously. Standard administration of the Decision Conflict Scale includes this item but it is not part of the DCS score.
Time Frame: Post test (2-3 weeks after pretest)
Population: Nursing Home Residents and Family Members
Measure: Number; unit: participants
Arm/Group | Decision Aid | No Decision Aid
Number analyzed (Participants) | 84 | 78
participants
  Prefer Hospital | 17 | 23
  Prefer Nursing Home | 17 | 6
  No Response | 50 | 49

5. Secondary Outcome: 30 Day Hospital Readmission
Description: Report of all hospitalizations from facility staff or participants Hospital Transfers Occurring During Study Period, i.e., number of resident participants who were hospitalized from pretest to posttest and by end of 3 month follow-up period.
Time Frame: Length of stay ≤30 days at Post test
Population: Nursing Home Residents and Family Members
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | No Decision Aid
Number analyzed (Participants) | 87 | 83
Participants | 8 | 5

ADVERSE EVENTS:
Time Frame: 6-8 months
Description: Serious adverse events reported to IRB
Arm/Group | Decision Aid | No Decision Aid
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/95
Other Adverse Events (participants affected / at risk) | 0/97 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No